CLINICAL TRIAL: NCT04540367
Title: Blood Flow Restriction Training for The Shoulder: A Case for Proximal Benefit
Brief Title: Blood Flow Restriction Training for The Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00017362
Record Dates: First submitted 2020-08-26; First posted 2020-09-07 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Healthy
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Participants were randomized to either perform exercises with blood flow restriction therapy or without
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- No Intervention: Control (No Intervention): Participants in this group performed the exercises without the blood flow restriction therapy cuff
- Experimental: BFR (Experimental): Participants in this group performed the exercises with the blood flow restriction therapy cuff
  Interventions: Device: Blood flow restriction therapy

INTERVENTIONS:
Device: Blood flow restriction therapy — The study group underwent the same exercises as the control group modified by the use of a tourniquet for blood flow restriction during those exercises.
  Arms: Experimental: BFR

SUMMARY:
The aim of this study is to determine if BFR-LIX promotes greater increases in shoulder lean mass, rotator cuff strength, endurance, and acute increases in shoulder muscle activation compared to LIX alone.

DETAILED DESCRIPTION:
Healthy Volunteers: Thirty-two healthy adults were randomized into two groups (BFRm=13,f=3, NoBFRm=10,f=6) that performed 8wks of shoulder LIX [2/wk, 4 sets (30/15/15/fatigue), 20%max] using common rotator cuff exercises [cable external rotation (ER), cable internal rotation (IR), dumbbell scaption (SCAP), and side-lying dumbbell ER (SLER)]. The BFR group also trained with an automated tourniquet placed at the proximal arm (50%-occlusion). Regional lean mass (dual-energy-xray-absorptiometry), isometric strength, and muscular endurance (repetitions-to-fatigue, RTF, 20%max, with and without 50%-occlusion) was measured before and after training. Electromyographic amplitude (EMGa) was also recorded from target shoulder muscles during endurance testing. A mixed-model ANCOVA (covaried on baseline measures) was used to detect within and between-group differences in primary outcome measures (α=0.05).

Pitchers: Twenty-eight collegiate baseball pitchers were randomized into 2 groups (BFRN=15, NOBFRN=13) that, in conjunction with offseason training, performed 8wks of shoulder LIX [Throwing arm only; 2/wk, 4 sets (30/15/15/fatigue), 20%isometric max] using 4 exercises [cable external and internal rotation (ER/IR), dumbbell scaption, and side-lying dumbbell ER]. The BFR group also trained with an automated tourniquet on the proximal arm (50%-occlusion). Regional lean mass (dual-energy x-ray absorptiometry), rotator cuff strength (dynamometry: IR0&90, ° ER0&90, ° Scaption, Flexion), and fastball biomechanics were assessed pre- and post-training. Achievable workload (sets × reps × resistance) was also recorded. An ANCOVA (covaried on baseline measures) repeated on training timepoint was used to detect within-group and between-group differences in outcome measures (α=0.05). For significant pairwise comparisons, effect size (ES) was calculated using a Cohen's d statistic and interpreted as: 0-0.1, negligible(N); 0.1-0.3, small(S); 0.3-0.5, moderate(M); 0.5-0.7, large(L); >0.7, very large(VL).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, untrained volunteers

Exclusion Criteria:

1. Previous history of shoulder injury occurring in the laterality of choice
2. Current painful dysfunction resulting in exercise limitation
3. Any health-related exercise limitation as ordered by physician
4. Vascular compromise or previous vascular surgery
5. Ages outside of 18-65
6. Inability to access clinic and equipment
7. Currently involved in structured strength training regimen of the upper extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick C McCulloch, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams GR. Invited Review: Autocrine/paracrine IGF-I and skeletal muscle adaptation. J Appl Physiol (1985). 2002 Sep;93(3):1159-67. doi: 10.1152/japplphysiol.01264.2001. PMID 12183514
- [Background] Burd NA, Holwerda AM, Selby KC, West DW, Staples AW, Cain NE, Cashaback JG, Potvin JR, Baker SK, Phillips SM. Resistance exercise volume affects myofibrillar protein synthesis and anabolic signalling molecule phosphorylation in young men. J Physiol. 2010 Aug 15;588(Pt 16):3119-30. doi: 10.1113/jphysiol.2010.192856. Epub 2010 Jun 25. PMID 20581041
- [Background] Cifrek M, Medved V, Tonkovic S, Ostojic S. Surface EMG based muscle fatigue evaluation in biomechanics. Clin Biomech (Bristol). 2009 May;24(4):327-40. doi: 10.1016/j.clinbiomech.2009.01.010. Epub 2009 Mar 13. PMID 19285766
- [Background] Cook SB, Clark BC, Ploutz-Snyder LL. Effects of exercise load and blood-flow restriction on skeletal muscle function. Med Sci Sports Exerc. 2007 Oct;39(10):1708-13. doi: 10.1249/mss.0b013e31812383d6. PMID 17909396
- [Background] Cools AM, De Wilde L, Van Tongel A, Ceyssens C, Ryckewaert R, Cambier DC. Measuring shoulder external and internal rotation strength and range of motion: comprehensive intra-rater and inter-rater reliability study of several testing protocols. J Shoulder Elbow Surg. 2014 Oct;23(10):1454-61. doi: 10.1016/j.jse.2014.01.006. Epub 2014 Apr 13. PMID 24726484
- [Background] Cools AM, Vanderstukken F, Vereecken F, Duprez M, Heyman K, Goethals N, Johansson F. Eccentric and isometric shoulder rotator cuff strength testing using a hand-held dynamometer: reference values for overhead athletes. Knee Surg Sports Traumatol Arthrosc. 2016 Dec;24(12):3838-3847. doi: 10.1007/s00167-015-3755-9. Epub 2015 Aug 21. PMID 26294055
- [Background] Cornish SM, Bugera EM, Duhamel TA, Peeler JD, Anderson JE. A focused review of myokines as a potential contributor to muscle hypertrophy from resistance-based exercise. Eur J Appl Physiol. 2020 May;120(5):941-959. doi: 10.1007/s00421-020-04337-1. Epub 2020 Mar 6. PMID 32144492
- [Background] Counts BR, Dankel SJ, Barnett BE, Kim D, Mouser JG, Allen KM, Thiebaud RS, Abe T, Bemben MG, Loenneke JP. Influence of relative blood flow restriction pressure on muscle activation and muscle adaptation. Muscle Nerve. 2016 Mar;53(3):438-45. doi: 10.1002/mus.24756. Epub 2015 Dec 29. PMID 26137897
- [Background] Dankel SJ, Jessee MB, Abe T, Loenneke JP. The Effects of Blood Flow Restriction on Upper-Body Musculature Located Distal and Proximal to Applied Pressure. Sports Med. 2016 Jan;46(1):23-33. doi: 10.1007/s40279-015-0407-7. PMID 26446893
- [Background] Figueiredo VC, de Salles BF, Trajano GS. Volume for Muscle Hypertrophy and Health Outcomes: The Most Effective Variable in Resistance Training. Sports Med. 2018 Mar;48(3):499-505. doi: 10.1007/s40279-017-0793-0. PMID 29022275
- [Background] Glowacki SP, Martin SE, Maurer A, Baek W, Green JS, Crouse SF. Effects of resistance, endurance, and concurrent exercise on training outcomes in men. Med Sci Sports Exerc. 2004 Dec;36(12):2119-27. doi: 10.1249/01.mss.0000147629.74832.52. PMID 15570149
- [Background] Hollman JH, Berling TA, Crum EO, Miller KM, Simmons BT, Youdas JW. Do Verbal and Tactile Cueing Selectively Alter Gluteus Maximus and Hamstring Recruitment During a Supine Bridging Exercise in Active Females? A Randomized Controlled Trial. J Sport Rehabil. 2018 Mar 1;27(2):138-143. doi: 10.1123/jsr.2016-0130. Epub 2018 Mar 1. PMID 28121207
- [Background] Hughes L, Paton B, Rosenblatt B, Gissane C, Patterson SD. Blood flow restriction training in clinical musculoskeletal rehabilitation: a systematic review and meta-analysis. Br J Sports Med. 2017 Jul;51(13):1003-1011. doi: 10.1136/bjsports-2016-097071. Epub 2017 Mar 4. PMID 28259850
- [Background] Hughes L, Rosenblatt B, Gissane C, Paton B, Patterson SD. Interface pressure, perceptual, and mean arterial pressure responses to different blood flow restriction systems. Scand J Med Sci Sports. 2018 Jul;28(7):1757-1765. doi: 10.1111/sms.13092. Epub 2018 Apr 30. PMID 29630752
- [Background] Illyes A, Kiss RM. Shoulder muscle activity during pushing, pulling, elevation and overhead throw. J Electromyogr Kinesiol. 2005 Jun;15(3):282-9. doi: 10.1016/j.jelekin.2004.10.005. PMID 15763675
- [Background] Lambert B, Hedt C, Epner E, et al. BFR For Proximal Benefit: Blood Flow Restriction Therapy For The Shoulder?: 3527: Board# 215 June 1 9: 30 AM-11: 00 AM. Med Sci Sports Exerc. 2019;51(6):972-973.
- [Background] Lambert B, Hedt CA, Jack RA, et al. Blood Flow Restriction Therapy Preserves Whole Limb Bone and Muscle Following ACL Reconstruction. Orthop J Sports Med. 2019;7(3_suppl2):2325967119S2325900196.
- [Background] Lambert BS, Hedt C, Moreno M, Harris JD, McCulloch P. Blood Flow Restriction Therapy for Stimulating Skeletal Muscle Growth: Practical Considerations for Maximizing Recovery in Clinical Rehabilitation Settings. Tech Orthop. 2018;33(2):89-97
- [Background] Lambert BS, Shimkus KL, Fluckey JD, Riechman SE, Greene NP, Cardin JM, Crouse SF. Anabolic responses to acute and chronic resistance exercise are enhanced when combined with aquatic treadmill exercise. Am J Physiol Endocrinol Metab. 2015 Feb 1;308(3):E192-200. doi: 10.1152/ajpendo.00689.2013. Epub 2014 Nov 25. PMID 25425002
- [Background] Loenneke JP, Kim D, Fahs CA, Thiebaud RS, Abe T, Larson RD, Bemben DA, Bemben MG. Effects of exercise with and without different degrees of blood flow restriction on torque and muscle activation. Muscle Nerve. 2015 May;51(5):713-21. doi: 10.1002/mus.24448. PMID 25187395
- [Background] Madarame H, Neya M, Ochi E, Nakazato K, Sato Y, Ishii N. Cross-transfer effects of resistance training with blood flow restriction. Med Sci Sports Exerc. 2008 Feb;40(2):258-63. doi: 10.1249/mss.0b013e31815c6d7e. PMID 18202577
- [Background] Mattocks KT, Jessee MB, Counts BR, Buckner SL, Grant Mouser J, Dankel SJ, Laurentino GC, Loenneke JP. The effects of upper body exercise across different levels of blood flow restriction on arterial occlusion pressure and perceptual responses. Physiol Behav. 2017 Mar 15;171:181-186. doi: 10.1016/j.physbeh.2017.01.015. Epub 2017 Jan 11. PMID 28088558
- [Background] Oishi Y, Tsukamoto H, Yokokawa T, Hirotsu K, Shimazu M, Uchida K, Tomi H, Higashida K, Iwanaka N, Hashimoto T. Mixed lactate and caffeine compound increases satellite cell activity and anabolic signals for muscle hypertrophy. J Appl Physiol (1985). 2015 Mar 15;118(6):742-9. doi: 10.1152/japplphysiol.00054.2014. Epub 2015 Jan 8. PMID 25571987
- [Background] Oliver JM, Kreutzer A, Jenke SC, Phillips MD, Mitchell JB, Jones MT. Velocity Drives Greater Power Observed During Back Squat Using Cluster Sets. J Strength Cond Res. 2016 Jan;30(1):235-43. doi: 10.1519/JSC.0000000000001023. PMID 26121432
- [Background] Paddon-Jones D, Sheffield-Moore M, Cree MG, Hewlings SJ, Aarsland A, Wolfe RR, Ferrando AA. Atrophy and impaired muscle protein synthesis during prolonged inactivity and stress. J Clin Endocrinol Metab. 2006 Dec;91(12):4836-41. doi: 10.1210/jc.2006-0651. Epub 2006 Sep 19. PMID 16984982
- [Background] Ploughman M, Shears J, Quinton S, Flight C, O'brien M, MacCallum P, Kirkland MC, Byrne JM. Therapists' cues influence lower limb muscle activation and kinematics during gait training in subacute stroke. Disabil Rehabil. 2018 Dec;40(26):3156-3163. doi: 10.1080/09638288.2017.1380720. Epub 2017 Oct 17. PMID 29041823
- [Background] Rome S, Forterre A, Mizgier ML, Bouzakri K. Skeletal Muscle-Released Extracellular Vesicles: State of the Art. Front Physiol. 2019 Aug 9;10:929. doi: 10.3389/fphys.2019.00929. eCollection 2019. PMID 31447684
- [Background] Salles JI, Velasques B, Cossich V, Nicoliche E, Ribeiro P, Amaral MV, Motta G. Strength training and shoulder proprioception. J Athl Train. 2015 Mar;50(3):277-80. doi: 10.4085/1062-6050-49.3.84. Epub 2015 Jan 16. PMID 25594912
- [Background] Sawilowsky SS. New effect size rules of thumb. J Mod Appl Stat Method. 2009;8(2):26.
- [Background] Scheuermann BW, Tripse McConnell JH, Barstow TJ. EMG and oxygen uptake responses during slow and fast ramp exercise in humans. Exp Physiol. 2002 Jan;87(1):91-100. doi: 10.1113/eph8702246. PMID 11805863
- [Background] Suga T, Okita K, Morita N, Yokota T, Hirabayashi K, Horiuchi M, Takada S, Omokawa M, Kinugawa S, Tsutsui H. Dose effect on intramuscular metabolic stress during low-intensity resistance exercise with blood flow restriction. J Appl Physiol (1985). 2010 Jun;108(6):1563-7. doi: 10.1152/japplphysiol.00504.2009. Epub 2010 Apr 1. PMID 20360434
- [Background] Suga T, Okita K, Takada S, Omokawa M, Kadoguchi T, Yokota T, Hirabayashi K, Takahashi M, Morita N, Horiuchi M, Kinugawa S, Tsutsui H. Effect of multiple set on intramuscular metabolic stress during low-intensity resistance exercise with blood flow restriction. Eur J Appl Physiol. 2012 Nov;112(11):3915-20. doi: 10.1007/s00421-012-2377-x. Epub 2012 Mar 14. PMID 22415101
- [Background] Takano H, Morita T, Iida H, Asada K, Kato M, Uno K, Hirose K, Matsumoto A, Takenaka K, Hirata Y, Eto F, Nagai R, Sato Y, Nakajima T. Hemodynamic and hormonal responses to a short-term low-intensity resistance exercise with the reduction of muscle blood flow. Eur J Appl Physiol. 2005 Sep;95(1):65-73. doi: 10.1007/s00421-005-1389-1. Epub 2005 Jun 15. PMID 15959798
- [Background] Takarada Y, Takazawa H, Ishii N. Applications of vascular occlusion diminish disuse atrophy of knee extensor muscles. Med Sci Sports Exerc. 2000 Dec;32(12):2035-9. doi: 10.1097/00005768-200012000-00011. PMID 11128848
- [Background] Takarada Y, Takazawa H, Sato Y, Takebayashi S, Tanaka Y, Ishii N. Effects of resistance exercise combined with moderate vascular occlusion on muscular function in humans. J Appl Physiol (1985). 2000 Jun;88(6):2097-106. doi: 10.1152/jappl.2000.88.6.2097. PMID 10846023
- [Background] Troiano A, Naddeo F, Sosso E, Camarota G, Merletti R, Mesin L. Assessment of force and fatigue in isometric contractions of the upper trapezius muscle by surface EMG signal and perceived exertion scale. Gait Posture. 2008 Aug;28(2):179-86. doi: 10.1016/j.gaitpost.2008.04.002. Epub 2008 May 19. PMID 18490165
- [Background] Yasuda T, Fujita S, Ogasawara R, Sato Y, Abe T. Effects of low-intensity bench press training with restricted arm muscle blood flow on chest muscle hypertrophy: a pilot study. Clin Physiol Funct Imaging. 2010 Sep;30(5):338-343. doi: 10.1111/j.1475-097X.2010.00949.x. Epub 2010 Jul 4. PMID 20618358

RESULTS

PARTICIPANT FLOW:
Groups:
- No Intervention: Control (General Population): Participants in this group performed the exercises without the blood flow restriction therapy cuff.
  Additionally, these participants are considered part of the general population.
- Experimental: BFR (General Population): Participants in this group performed the exercises with the blood flow restriction therapy cuff
  Blood flow restriction therapy: The study group underwent the same exercises as the control group modified by the use of a tourniquet for blood flow restriction during those exercises.
  Additionally, these participants are considered part of the general population.
- No Intervention: Control (Pitchers): Participants in this group performed the exercises without the blood flow restriction therapy cuff.
  Additionally, these participants are considered the pitchers.
- Experimental: BFR (Pitchers): Participants in this group performed the exercises with the blood flow restriction therapy cuff
  Blood flow restriction therapy: The study group underwent the same exercises as the control group modified by the use of a tourniquet for blood flow restriction during those exercises.
  Additionally, these participants are considered the pitchers.
Period: Overall Study
Arm/Group | No Intervention: Control (General Population) | Experimental: BFR (General Population) | No Intervention: Control (Pitchers) | Experimental: BFR (Pitchers)
Started | 16 | 16 | 18 | 19
Completed | 16 | 16 | 13 | 15
Not Completed | 0 | 0 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2
Not completed — COVID-19 Contact Tracing Protocols prevented completion of study activities | 0 | 0 | 4 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Intervention: Control (General Population) | Experimental: BFR (General Population) | No Intervention: Control (Pitchers) | Experimental: BFR (Pitchers) | Total
Number analyzed (Participants) | 16 | 16 | 13 | 15 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 13 | 15 | 60
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (8.3) | 27.6 (8.8) | 19.8 (1.5) | 19.7 (1.2) | 26.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 0 | 0 | 9
  Male | 10 | 13 | 13 | 15 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 13 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Determine if BFR Changes UE Lean Muscle Mass in the General Population
Description: UE lean muscle mass was measured in grams using DEXA. These data are reported as an average of both the left and right side.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: g
Groups:
- General Population, No Intervention: Control: Participants in this group performed the exercises without the blood flow restriction therapy cuff
- General Population, Experimental: BFR: Participants in this group performed the exercises with the blood flow restriction therapy cuff
  Blood flow restriction therapy: The study group underwent the same exercises as the control group modified by the use of a tourniquet for blood flow restriction during those exercises.
Arm/Group | General Population, No Intervention: Control | General Population, Experimental: BFR
Number analyzed (Participants) | 16 | 16
g
  Upper extremity lean muscle mass at 8 weeks | -17 (77) | 175 (54)
  Shoulder region lean muscle mass at 8 weeks | 96 (61) | 278 (90)

2. Primary Outcome: Isometric Rotator Cuff Strength in General Population
Description: Peak strength was measured using a hand-held dynamometer. A standardized procedure was used for shoulder strength testing, and all testing was performed by a sports-specialized (American Board of Physical Therapy Specialties Sports Clinical Specialist) physical therapist. A total of 6 different maximal isometric strength tests were used to measure the strength of the rotator cuff muscles in the following order: (1) seated forward flexion at 90 of shoulder abduction, (2) seated scaption at 90, (3) seated external rotation (ER) at 0, (4) seated internal rotation (IR) at 0, (5) prone ER at 90, and (6) prone IR at 90. Peak strength was measured using a microFET2 (Hoggan Scientific) hand-held dynamometer. For each isometric test, participants performed a 3-second maximal-exertion contraction against the dynamometer to determine peak strength. For each measure, tests were performed 3 times, and the highest value among the 3 trials was selected as the maximal strength value.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | No Intervention: Control | Experimental: BFR
Number analyzed (Participants) | 16 | 16
kg
  Pre Flexion | 12.1 (0.4) | 12.2 (0.4)
  Post Flexion | 11.9 (0.4) | 12.8 (0.4)
  Pre Scaption | 12 (0.2) | 12.1 (0.2)
  Post Scaption | 12.5 (0.2) | 12.4 (0.2)
  Pre ER at 0 | 13.7 (0.4) | 13.9 (0.4)
  Post ER at 0 | 13.9 (0.4) | 14.1 (0.4)
  Pre IR at 0 | 20.1 (0.7) | 20.2 (0.7)
  Post IR at 0 | 20.2 (0.7) | 23.1 (0.7)
  Pre ER at 90 | 15.6 (0.7) | 16 (0.7)
  Post ER at 90 | 14.7 (0.8) | 16.1 (0.7)
  Pre IR at 90 | 17.4 (0.8) | 17.9 (0.8)
  Post IR at 90 | 18.1 (0.8) | 18.6 (0.8)

3. Primary Outcome: Determine if BFR Changes Shoulder Lean Muscle Mass in Pitchers
Description: Shoulder lean muscle mass was measured in grams using DEXA. These data are reported for each arm.
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: g
Groups:
- Pitchers, No Intervention: Control: Participants in this group performed the exercises without the blood flow restriction therapy cuff
- Pitchers, Experimental: BFR: Participants in this group performed the exercises with the blood flow restriction therapy cuff
  Blood flow restriction therapy: The study group underwent the same exercises as the control group modified by the use of a tourniquet for blood flow restriction during those exercises.
Arm/Group | Pitchers, No Intervention: Control | Pitchers, Experimental: BFR
Number analyzed (Participants) | 13 | 15
g
  Shoulder Lean Muscle Mass in Throwing Arm at Baseline | 4291.8 (51.7) | 4279 (52)
  Shoulder Lean Muscle Mass in Non-Throwing Arm at Baseline | 4284.1 (55.9) | 4272.1 (55.5)
  Shoulder Lean Muscle Mass in Throwing Arm at 8 Weeks | 4307.3 (51.7) | 4410.1 (52)
  Shoulder Lean Muscle Mass in Non-Throwing Arm at 8 Weeks | 4347.3 (56) | 4346.2 (55.5)

4. Primary Outcome: Isometric Rotator Cuff Strength in Pitchers
Description: as for outcome 2
Time Frame: Baseline, 8 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Pitchers, No Intervention: Control | Pitchers, Experimental: BFR
Number analyzed (Participants) | 13 | 15
kg
  Pre Flexion in Throwing Arm | 14.8 (0.6) | 14.7 (0.5)
  Post Flexion in Throwing Arm | 13.2 (0.6) | 14.0 (0.5)
  Pre Flexion in Non-throwing arm | 14.7 (0.6) | 14.6 (0.5)
  Post flexion in Non-Throwing Arm | 14.2 (0.6) | 14.0 (0.5)
  Pre Scaption in Throwing Arm | 14.7 (0.6) | 14.7 (0.5)
  Post Scaption in Throwing Arm | 14.5 (0.6) | 14.5 (0.5)
  Pre Scaption in Non-Throwing Arm | 14.7 (0.6) | 14.7 (0.5)
  Post Scaption in Non-Throwing Arm | 14.1 (0.6) | 14.3 (0.5)
  Pre ER at 0 in Throwing Arm | 16.2 (0.9) | 15.9 (0.8)
  Post ER at 0 in Throwing Arm | 16.4 (0.9) | 15.8 (0.8)
  Pre ER at 0 in Non-Throwing Arm | 16.0 (0.9) | 16.0 (0.8)
  Post ER at 0 in Non-Throwing Arm | 16.0 (0.9) | 15.9 (0.8)
  Pre IR at 0 in Throwing Arm | 24.8 (1.4) | 24.3 (1.2)
  Post IR at 0 in Throwing Arm | 21.8 (1.4) | 25.4 (1.2)
  Pre IR at 0 in Non-Throwing Arm | 24.2 (1.3) | 24.1 (1.2)
  Post IR at 0 in Non-Throwing Arm | 22.5 (1.3) | 24.4 (1.2)
  Pre ER at 90 in Throwing Arm | 19.7 (1.4) | 19.7 (1.3)
  Post ER at 90 in Throwing Arm | 18.9 (1.4) | 17.3 (1.3)
  Pre ER at 90 in Non-Throwing Arm | 20.1 (1.4) | 20.0 (1.3)
  Post ER at 90 in Non-Throwing Arm | 21.1 (1.4) | 17.8 (1.3)
  Pre IR at 90 in Throwing Arm | 20.0 (1.5) | 19.7 (1.3)
  Post IR at 90 in Throwing Arm | 20.9 (1.5) | 22.1 (1.3)
  Pre IR at 90 in Non-Throwing Arm | 19.5 (1.5) | 19.9 (1.4)
  Post IR at 90 in Non-Throwing Arm | 21.4 (1.5) | 20.4 (1.4)

5. Secondary Outcome: Strength Endurance in General Population
Description: repetitions to fatigue (RTF) were performed for 3 exercises. Volume (repetitions x resistance, kg) was calculated for each trial as is common for strength training investigations.
  After strength testing, participants were asked to perform the first of 2 endurance tests separated by 48 to 72 hours. On both occasions, a single set of repetitions to fatigue (RTF) were performed for 3 exercises in the following order: standing cable ER at 0 of shoulder abduction, standing cable IR at 0, and dumbbell scaption with each exercise separated by a 2-minute rest period and alternating between arms (order randomized). This test was performed in both groups with and without 50% limb occlusion pressure (LOP) applied by an automated tourniquet system. A nylon cuff was placed around the most proximal portion of the upper extremity for all testing. The order of testing was randomized between the 2 testing days for each participant.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | No Intervention: Control | Experimental: BFR
Number analyzed (Participants) | 16 | 16
kg
  Cable ER - Pre at 50% LOP | 97.3 (10.8) | 94.1 (10.9)
  Cable ER Post at 50% LOP | 155.1 (10.8) | 155.1 (10.9)
  Cable IR - Pre at 50% LOP | 230.7 (19.5) | 230.9 (19.5)
  Cable IR - Post at 50% LOP | 305.9 (19.5) | 389.5 (19.6)
  Scaption - Pre at 50% LOP | 134.8 (18.8) | 137 (18.9)
  Scaption - Post at 50% LOP | 211.2 (18.8) | 240.3 (18.8)
  Cable ER - Pre without LOP | 99.5 (12.8) | 96.2 (10.8)
  Cable ER Post without LOP | 157.2 (10.7) | 155.9 (10.8)
  Cable IR - Pre at without LOP | 249.1 (17.8) | 249.3 (17.9)
  Cable IR - Post at without LOP | 342.2 (17.8) | 407 (17.9)
  Scaption - Pre at without LOP | 138.6 (18.3) | 140.2 (18.4)
  Scaption - Post without LOP | 222.7 (18.4) | 231.7 (18.4)

ADVERSE EVENTS:
Time Frame: The AE was a single episode of a muscle strain. The subject was monitored from the time of the event through study completion, an average of 8 weeks.
Description: It was a muscle strain as the volunteer had an untrained arm. It was treated with ibuprofen, the subject was completely fine and able to finish the study.
Arm/Group | No Intervention: Control (General Population) | Experimental: BFR (General Population) | No Intervention: Control (Pitchers) | Experimental: BFR (Pitchers)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/16 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/13 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | No Intervention: Control (General Population) (N=16) | Experimental: BFR (General Population) (N=16) | No Intervention: Control (Pitchers) (N=13) | Experimental: BFR (Pitchers) (N=15)
Other (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — The subject had an arm muscle strain from having an untrained arm. They were treated with ibuprofen, cleared by the PI and were able to complete the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT04540367/Prot_SAP_003.pdf